CLINICAL TRIAL: NCT04765501
Title: Cross-cultural Adaptation, Reliability and Validity of the Turkish Version of the Headache Impact Questionnaire
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: 83116987-555
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2022-10

CONDITIONS: Headache; Headache Disorders; Headache, Migraine; Headache, Tension; Headaches Chronic; Headaches Muscular
Keywords: Headache; Reliability; Validity; Cross-cultural adaptation
MeSH Terms: conditions — Headache; Headache Disorders; Migraine Disorders; Tension-Type Headache | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients group: Individuals with headache
  Interventions: Other: Survey study

INTERVENTIONS:
Other: Survey study — Headache Impact Questionnaire (HIQ) will be applied.

SUMMARY:
The purpose of this study was to investigate cultural adaptation, reliability and validity of the Turkish version of the Headache Impact Questionnaire (HIQ).

DETAILED DESCRIPTION:
The episodic nature of migraine attacks presents a number of difficulties in characterizing disease severity. There are differences in the severity, frequency and intensity of attacks and the general effect of the disease in individuals. Information about any particular attack is not sufficient to characterize the overall severity of the disease. Accordingly, the Headache Impact Questionnaire (HIQ) was developed to evaluate the headache experience over a period of time instead of any headache. Developed to measure the impact and quality of life of individuals suffering from headache, hıq evaluates the frequency and duration of headache, the degree of pain severity, daily life activities, disruptions in work or school life, the influence of the individual's leisure activities and other symptoms that may occur. HIQ consists of 16 items and the higher the score shows the seriousness of the impact. The study is planned with 80 individuals with complaint of headache. After questioning the sociodemographic characteristics of the individuals, the patients will be asked to fill in HIQ, Migraine Disability Assessment Questionnaire, Headache Impact Test-6 and Short Form-36.Test-retest will be re-applied to those of the same individuals who can be reached after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any type of headache,
* Have a chronic headache.

Exclusion Criteria:

* Having a cognitive and neurological disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with any type of headache.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Headache Impact Questionnaire (HIQ) | 15 minutes
  Headache Impact Questionnaire is designed to measure the quality of life related to the disability

CONTACTS AND LOCATIONS:
Locations (1):
- Halime ARIKAN, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR